CLINICAL TRIAL: NCT05207982
Title: Weight Management Program for Patients With First Episode Psychosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Daniel Antonius, Associate Professor, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Antonius (Pilot 2022); UL1TR001412 (NIH)
Record Dates: First submitted 2022-01-04; First posted 2022-01-26 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Diet, Healthy; Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Family Based weight management program — Weight management program that involve the patient AND a family member or a care taker. Families will receive a 12-week FBT adapted for first episode psychosis. This will be delivered in 12 weekly meetings with a trained case manager and two "eating plan" education sessions. Both the patient with psychosis and parents are targeted for eating and activity/exercise change to ensure a change in the shared family environment, which will also help weight control in both sets of participants, as well as medical issues that accompany obesity, including glycemic control, hypertension and hyperlipidemia. If parents are not overweight/obese, they will still target improved health behaviors. They will learn about GREEN, YELLOW, and RED foods (healthy vs. unhealthy foods), energy density, glycemic index of foods, reducing serving sizes, eating less, healthy lifestyle and programmed activity programs and recording their diets and activity.

SUMMARY:
Severe mental illnesses (SMI), such as schizophrenia, are associated with increased morbidity and mortality in large part due to obesity and concomitant metabolic disorders. People with SMI have twice the risk of becoming obese, driven by the use of antipsychotic medications. These antipsychotic medications are dopamine antagonists, which reduce brain dopamine levels, leading to an increase in food reinforcement, which leads to weight gain. This weight gain occurs very rapidly with the initiation of these medications, as do increases in LDL cholesterol, insulin, and leptin.

While there have been attempts to develop weight loss programs, a recent meta-analysis concluded that these interventions led to statistically significant weight loss that was of no clinical significance and did not last beyond the intervention. Given the rapid weight gain/metabolic changes and the findings that it is easier to prevent weight gain than to lose weight, interventions targeting the early phases of a first episode of psychosis (FEP) are critical. However, the very few attempts have failed to address two key aspects of first episode psychosis. First, antipsychotic medications increase the reinforcing value of food and interventions have not included strategies to provide alternative reinforcements. Second, most patients experiencing FEP live with and are dependent on their parents, but existing interventions have not utilized parents in support of exercise and dietary changes.

The purpose of this project is to assess the feasibility and acceptability of, and to provide preliminary evidence for the efficacy of a Family-Based Treatment (FBT) that includes both the patient and the parent in the intervention and provides structured help in developing alternative reinforcements that support exercise and dietary changes. The specific aims of this project are:

1. Recruit and provide FBT to 12 FEP patients and their parents using a multiple baseline single case experimental design;
2. Evaluate participation, attrition, and satisfaction of the patients and their families across the three month treatment period;
3. Examine the hypothesis that weight and food reinforcement will be significantly reduced during the treatment and follow-up phases in contrast to the baseline period.

DETAILED DESCRIPTION:
C. Overview Study Sample: Twelve families will be recruited from NAVIGATE, a program for first episode psychosis patients. Patients in the program and who have been prescribed antipsychotic medications will be eligible. In addition, to be eligible, one of the parents must agree to work with the patient, and agree to modify their eating, exercise and if obese, their own weight. Patients and parents must be able to read at the 8th grade level. Patients or parents with a history or evidence of current eating disorders (bulimia or anorexia or binge eating disorder) or a current alcohol or drug use disorder will be excluded.

The NAVIGATE program admits 2 to 3 patients per month. At the beginning of the study, we anticipate that there would be approximately 40-45 patients in the program with the requisite use of antipsychotic medications, and over the next five months, we would expect an additional 10-15 patients. Assuming that 50% of the patients are eligible and interested, we would have approximately 25-30 patients available for the study.

Assessments: Participants will have a baseline session in which they complete the Behavioral Choice Questionnaire that assesses the reinforcing value of food. Parents and the patients will also complete questionnaires regarding parenting, time perspective, consideration of future consequences, and have their height and weight measured. Following the baseline assessment, baseline data will be collected over a two month period, and then families will be randomized to staggered initiation of treatment in blocks of 4 families. At the end of treatment, the patient and the participating parent will receive the same assessment battery that they completed for the baseline session. They will also provide information on the implementation of the diet, exercise, and alternative reinforcement procedures. After an additional 2 months, the patient and parent will return for the final assessment using the same assessment battery, as well as the implementation data.

During the baseline, treatment and follow-up period, patients will take their weight daily with a Bluetooth scale provided by the project.

Intervention: Families will receive a 12-week FBT adapted for first episode psychosis. This will be delivered in 12 weekly meetings with a trained case manager and two "eating plan" education sessions. Both the patient with psychosis and parents are targeted for eating and activity/exercise change to ensure a change in the shared family environment, which will also help weight control in both sets of participants, as well as medical issues that accompany obesity, including glycemic control, hypertension and hyperlipidemia. If parents are not overweight/obese, they will still target improved health behaviors. They will learn about GREEN, YELLOW, and RED foods (healthy vs. unhealthy foods), energy density, glycemic index of foods, reducing serving sizes, eating less, healthy lifestyle and programmed activity programs and recording their diets and activity. Weekly sessions will involve discussion of weight loss principles presented in modules in the weight control manual, and coaching parents and patients how to implement the Traffic Light Eating Plan and healthy lifestyle techniques. At each session, participants meet with staff and attend a brief problem solving session with their case manager where they will troubleshoot any expected or encountered issues with implementing the program. As part of treatment, participants will weigh themselves daily with a Bluetooth scale.

An innovative aspect of this treatment is helping patients develop alternative reinforcements that do not involve food that can reduce the motivation to eat for the hedonic or reinforcing motivations. The first step is to identify alternative activities that have a higher reinforcement value than the patients' favorite foods. First, participants will identify potential alternatives from the 139 behaviors on the Pleasant Activities List. The therapist then works with the patient to better specify the behavior, ensure its feasibility and describe the parameters of the behavior (e.g. duration). After the participant and case manager agree on a list of alternatives (at least 5), the participant will complete the Behavioral Choice Questionnaire that assesses the reinforcing value of that activity in comparison to food. The most reinforcing food to be used to assess behavioral substitutes will be chosen from a list of usual meals that can be obtained from home cooked, fast food or casual dining restaurants. These alternative reinforcements are used non-contingently by the patients/parents to provide highly desirable activities that compete with excessive food consumption.

Design and analysis: The project is a multiple baseline single case experimental design, with a 2 month baseline data collection. Families will then be randomized to staggered initiation of treatment in blocks of 4 families. We anticipate having 8 participating families at the beginning of the project and would randomly assign them to start the baseline assessment between 1 and 9 weeks into the project, with the treatment then beginning between weeks 9 and 17. Treatment completion for this initial cohort would be between weeks 21 and 29, and the final follow-up would occur between weeks 29 and 37. Families entering NAVIGATE after the recruitment of the first cohort will be randomly assigned to start the baseline from 1 to 9 weeks after entry. This will provide a significant baseline (2 months) for all participants with different initial points for the study.

Analysis of the daily weights will involve discontinuous growth curve analysis using multi-level modeling. Separate models are developed for each participant which include the daily weights from the baseline (60 days), treatment (90 days) and follow-up (60 days) phases. Given the nature of the data, we would hypothesize significantly different slopes for the baseline vs treatment phases. We would also expect no significant differences between the slopes for the treatment phase and the follow-up phase. The primary analysis involves modeling each individual as a level one variable. This data may be examined at the individual level to provide information regarding the number of individuals responding to the treatment, as well as through meta-analysis to provide more specific effect sizes.

ELIGIBILITY:
Inclusion Criteria:

Participant:

* Age 14-26 years
* Enrolled in NAVIGATE, a clinical program for patients with first episode of psychosis.
* Prescribed antipsychotic medication for a first break psychotic episode
* Availability of household family member to collaborate in the weight management program.

Family Member:

* Lives in the same household as participant (e.g., parent, guardian, grandparent, aunt or uncle)
* Able to attend weekly meetings with a case manager

Exclusion Criteria:

Participant & Family Member:

* Personal or Family history or evidence of current eating disorders (bulimia or anorexia or binge eating disorder)
* Current alcohol or drug abuse,
* Unable to read at 8th grade level
* Unable to use technology.
* Unable to weigh themselves daily due to existing medical condition
* Pregnant or planning on becoming pregnant during the study

Ages: 14 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Erie County Medical Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McElroy SL. Obesity in patients with severe mental illness: overview and management. J Clin Psychiatry. 2009;70 Suppl 3:12-21. doi: 10.4088/JCP.7075su1c.03. PMID 19570497
- [Background] Gates J, Killackey E, Phillips L, Alvarez-Jimenez M. Mental health starts with physical health: current status and future directions of non-pharmacological interventions to improve physical health in first-episode psychosis. Lancet Psychiatry. 2015 Aug;2(8):726-742. doi: 10.1016/S2215-0366(15)00213-8. PMID 26249304
- [Background] Daurignac E, Leonard KE, Dubovsky SL. Increased lean body mass as an early indicator of olanzapine-induced weight gain in healthy men. Int Clin Psychopharmacol. 2015 Jan;30(1):23-8. doi: 10.1097/YIC.0000000000000052. PMID 25350366
- [Background] Tek C, Kucukgoncu S, Guloksuz S, Woods SW, Srihari VH, Annamalai A. Antipsychotic-induced weight gain in first-episode psychosis patients: a meta-analysis of differential effects of antipsychotic medications. Early Interv Psychiatry. 2016 Jun;10(3):193-202. doi: 10.1111/eip.12251. Epub 2015 May 12. PMID 25962699
- [Background] Epstein LH, Bickel WK, Czajkowski SM, Paluch RA, Moeyaert M, Davidson KW. Single case designs for early phase behavioral translational research in health psychology. Health Psychol. 2021 Dec;40(12):858-874. doi: 10.1037/hea0001055. Epub 2021 Aug 9. PMID 34370494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dyads consisting of patients and their support person (one patient and one support person per dyad) were recruited from an outpatient clinic between 7/15/22 and 6/30/23
Groups:
- Patients: Patients with first episode psychosis (FEP) participating in the weight management program
- Supporting Person: Supporting person assisting the FEP patient in the weight management program
Period: Overall Study
Arm/Group | Patients | Supporting Person
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients | Supporting Person | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (3.1) | 38.2 (15.5) | 30 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Weight [Mean (Full Range); unit: Lbs] — Daily weights from participants collected via Bluetooth scales
  Lbs | 217.3 [190.9 to 239.2] | 201.5 [150.6 to 236.3] | 209.4 [150.6 to 239.2]

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Change in weight will be assessed at baseline, weekly during study period, end point, and follow up.
Time Frame: 7 months
Population: This is a single case experimental, within-subject, design study, in which participants' weight at baseline and after intervention is being measured. Separate models were used for each participant and total weight loss (number) were examined.
Measure: Number; unit: Lbs
Arm/Group | Patients | Supporting Person
Number analyzed (Participants) | 5 | 5
Lbs
  Dyad 1: number analyzed (Participants) | 1 | 1
  Dyad 1 | -6 | -3
  Dyad 2: number analyzed (Participants) | 1 | 1
  Dyad 2 | -5 | -4
  Dyad 3: number analyzed (Participants) | 1 | 1
  Dyad 3 | 11 | 5
  Dyad 4: number analyzed (Participants) | 1 | 1
  Dyad 4 | -4 | -14
  Dyad 5: number analyzed (Participants) | 1 | 1
  Dyad 5 | 0 | -7
Statistical Analysis 1: Comparison: Patients vs Supporting Person; This study utilized a multiple baseline single case experimental design in which analysis of the daily weights (for each participant) involved discontinuous growth curve analysis using multi-level modeling. Separate models were developed for each participant which include the daily weights from the baseline, treatment and follow-up phases. Given the nature of the data, we hypothesized different slopes for the baseline vs treatment phases. Overall weight change was a primary outcome measure; Test type: Other; Multiple baseline single case experimental design in which analysis of the daily weights (for each participant) involved discontinuous growth curve analysis using multi-level modeling

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Patients | Supporting Person
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT05207982/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT05207982/ICF_001.pdf